CLINICAL TRIAL: NCT06316232
Title: Efficacy of Deep Brain Stimulation and Levodopa on Freezing of Gait in Advanced Parkinson's Disease: a Comparative Study
Brief Title: DBS and Levodopa for Treating Freezing of Gait in Parkinson's Disease
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS Istituto delle Scienze Neurologiche di Bologna (Other)
Collaborators: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Ilaria Cani, Principal Investigator, IRCCS Istituto delle Scienze Neurologiche di Bologna
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DBS-FOG 2023
Record Dates: First submitted 2024-03-01; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Freezing of Gait; Parkinson Disease
Keywords: freezing of gait; gait disturbances; parkinson disease
MeSH Terms: conditions — Parkinson Disease; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: In addition to baseline gait assessment performed in a morning session on MED ON/STIM ON condition (after usual levodopa morning dose and usual parameters of stimulation), patients are evaluated in two following morning sessions under different treatment conditions:
  1. STIM ON plus: evaluation after the administration of levodopa morning dose and the increase of intensity of stimulation of 0.5 mA bilaterally,
  2. MED ON plus: evaluation after the administration of a 2x levodopa morning dose with usual parameters of stimulation.
Who Masked: Outcomes Assessor
Masking Description: The count and duration of FoG episodes during the standardize walking protocol is measured on video-assessment by two blind raters.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STIM ON plus/MED ON plus (Active Comparator): Patients were evaluated in two following morning sessions under different treatment conditions:
  1. STIM ON plus (intervention 1)
  2. MED ON plus (intervention 2)
  Interventions: Device: STIM ON plus; Drug: MED ON plus
- MED ON plus/STIM ON plus (Active Comparator): Patients were evaluated in two following morning sessions under different treatment conditions:
  1. MED ON plus (intervention 2)
  2. STIM ON plus (intervention 1)
  Interventions: Device: STIM ON plus; Drug: MED ON plus

INTERVENTIONS:
Device: STIM ON plus — increase of intensity of stimulation of 0.5 mA bilaterally
Drug: MED ON plus — administration of a 2x levodopa morning dose

SUMMARY:
Freezing of gait (FoG) is a complex symptom of Parkinson's disease (PD) that cause falls and disability in PD patients, heavily affect patients' autonomy and quality of life. Gait disturbances and FoG are difficult to manage as they usually do not complete respond to both dopaminergic treatment and subthalamic nucleus deep brain stimulation (STN-DBS). One therapeutic strategy suggested in literature for improving gait disturbances is to increase the dose of dopaminergic drugs according to the hypothesis of pseudo-ON-freezing. The pseudo-ON-FoG in patients treated with STN-DBS can easily occur as the result of a suboptimal stimulation or the consequence of a post-operative reduction of the dopaminergic therapy. Therefore, it is reasonable hypothesize both the increase of stimulation and levodopa as good therapeutic strategies to improve pseudo-ON-FoG. At present there are no evidence for suppose that one option is better than the other, even though two recent studies on gait analysis reported a positive additive effect of levodopa therapy on gait parameters in patients treated with STN-DBS.

In this study, the investigators aim to objectively evaluating the improvement of FoG in PD patients treated with STN-DBS at different treatment conditions consisting of increased intensity of stimulation or higher dosage of levodopa.

DETAILED DESCRIPTION:
This is a cross-over, blind, randomized study to evaluate the improvement of FoG in a group of PD patients treated with bilateral STN-DBS by increasing the intensity of stimulation (STIM plus) or administering a higher dose of levodopa (MED plus).

Patient will be videorecorded for evaluation of freezing episodes and gait cinematic parameters by means of 3 wearable inertial sensors on the feet and at lumbar level during a standardized walking protocol including: Timed Up and Go, Turn 360°, Gait 18 m and a Complex task in single task and dual task (serial-3 subtractions) conditions. In each condition, Tinetti scale, Trail Making Test, alternate fluency test, Movement Disorders Society Unified Parkinson's disease Rating Scale (MDS-UPDRS) and MDS Unified Dyskinesia Rating Scale (UDysRS) will be also perform.

In addition, other demographic and clinical information such as age, sex, MMSE, MoCA, New Freezing of Gait Questionnaire, Falls Efficacy Scale will be collected.

The primary endpoint of this study is to investigate the efficacy of increasing intensity of stimulation (STIM plus) or levodopa (MED plus) on freezing of gait (FOG).

Secondary outcome measures include cinematic gait parameters, global motor outcomes and cognitive functions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's disease treated with STN-DBS who achieved a good control of motor fluctuations and cardinal motor symptoms (bradykinesia, rigidity, tremor)
* History of FoG in daily-ON condition after optimal DBS programming, defined by a score of 1 on Question 1 and score ≥ 2 on Question 2 of the New Freezing of Gait Questionnaire.

Exclusion Criteria:

* inability to walk independently for 10 meters.
* limited therapeutic windows of stimulation without the possibility of increase the intensity of stimulation of 0,5 mA for the appearance of side effects
* previous evidence of severe adverse effects with high levodopa dose ore increased STN-DBS intensity, such as psychosis, hallucinations, painful dyskinesias, severe hypotension, digestive symptoms.
* dementia (MMSE score ≤ 18)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Time spent with FOG during protocol | immediate post monitoring
  Video-assessed reduction in the total time of FoG during the standardize walking protocol in MED ON plus or STIM ON plus condition compared to baseline.

SECONDARY OUTCOMES:
Gait performance | immediate post monitoring
  Changes in gait parameters measured by a system of 3 wearable inertial sensors, including: gait speed, stride lenght, number of step, cadence, gait variability, left-right asymmetry during MED ON plus or STIM ON plus protocol compared to baseline.
MDS-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III | immediate post monitoring
  Change in items 3.10 and 3.11 MDS UPDRS part III and total score between MED ON plus or STIM ON plus condition and baseline.
Patient global impression of change (PGI-C) | immediate post monitoring
  Change in PGI-C scores on MED ON plus or STIM ON plus condition compared to baseline.
Trail Making test A and B | immediate post monitoring
  Change in Trail Making test A and B scores during MED ON plus or STIM ON plus protocol compared to baseline.
Phonemic/Semantic alternate Fluency test | immediate post monitoring
  Change in during Phonemic/Semantic alternate Fluency test scores between MED ON plus or STIM ON plus condition and baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Ilaria Cani, Principal Investigator — IRCCS Istituto delle Scienze Neurologiche di Bologna
Locations (1):
- IRCCS Istituto delle Scienze Neurologiche di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No